CLINICAL TRIAL: NCT05941546
Title: Tick-borne Encephalitis Virus Research in Limousin
Acronym: VITAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI23_0012
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Tick-borne Encephalitis
Keywords: tick-borne encephalitis; TBEV; serology; PCR
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: anti-TBEV serology — we will measure by ELISA in microplates the anti-TBEV IgG as well as the anti-TBEV IgM on the sera + in TBEV IgG. We will then send a patient questionnaire with an information note to document the context of this TBEV seropositivity and to eliminate false-positivities (vaccination). Finally, we will perform PCR on CSF if serum positive and CSF available

SUMMARY:
Cases of encephalitis of varying severity have been described in recent years in eastern France involving tick-borne encephalitis virus (TBEV). The main objective is to demonstrate the presence of TBEV in Limousin, in patients with a positive Lyme serology, or a neurological picture compatible with TBEV.

DETAILED DESCRIPTION:
Cases of encephalitis of varying severity have been described in recent years in eastern France involving tick-borne encephalitis virus (TBEV). The epidemiological situation in France is poorly known with about 20 cases diagnosed per year, mainly in Alsace and Haute-Savoie. The infection can result in fever and an influenza-like picture, which can be complicated by encephalitis-like neurological disorders, or even death. TBEV is transmitted by the tick Ixodes ricinus, which also carries Borrelia burgdorferi, the agent of Lyme disease. Limousin is one of the French regions with the highest prevalence of Lyme disease. These ticks can harbor various pathogens, including TBEV. A case was described in 2007 in Bordeaux. More recently, a case was described in Haute-Loire. The investigators are therefore interested today in the emergence of this virus in Limousin following a possible progression through the Massif Central, potentially favored by numerous anti-Covid-19 control containments. The study begins with a computer extraction of patients with Lyme serology from our GLIMS laboratory software (with positive or negative results), a check for non-oppositions. Then the investigators will measure by ELISA in microplates the anti-TBEV IgG as well as the anti-TBEV IgM on the sera + in TBEV IgG. The investigators will then send a patient questionnaire with an information note to document the context of this TBEV seropositivity and to eliminate false-positivities (vaccination). Finally, the investigators will perform PCR on CSF if serum positive and CSF available, followed by an analysis of results.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Lyme serology. Neurological picture compatible with neuroborreliosis or encephalitis.
* No objection from the patient to the use of biobank samples

Exclusion Criteria:

* Patient's opposition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with Lyme serology from our GLIMS laboratory software (with positive or negative results)
Sampling Method: Non-Probability Sample
Enrollment: 878 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-08-13 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
Detection of anti-TBEV antibodies in serum | month 1
  The primary endpoint is the detection of anti-TBEV antibodies in the serum of the study population.

SECONDARY OUTCOMES:
Search for the presence of TBEV in the CSF in case of positive serology. Determine the risk factors associated with this infection. | month 2
  the detection of TBEV RNA will be carried out by real-time RT-PCR in the CSF of patients with positive anti-TBEV serology (if associated CSF available). The analysis will be qualitative in order to obtain a positive/negative response on the presence of virus RNA in the sample.
  In order to obtain information on the context of the infection, a questionnaire will be sent to TBEV-positive patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hosiptal, Limoges, France

IPD SHARING:
Plan to Share IPD: No